CLINICAL TRIAL: NCT04533321
Title: A Biomarker-implemented Clinical Study Evaluating Mutations in MET and TP53 in a Population of Treatment-refractory Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC01/02/20
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Squamous Cell Carcinoma
Keywords: MET; TP53
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients genotyped positive for MET-N375S polymorphism (Other): will be treated with orally administered daily dose of afatinib (Gilotrif®) in a fasting state (1 hour before or 2 hours after meals).
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Afatinib is approved therapy for SCC of the lung after progression with standard of care chemotherapy.

SUMMARY:
Afatinib is approved therapy for SCC of the lung after progression with standard of care chemotherapy. There is also evidence of improvement of progression free survival of patients with metastatic/recurrent SCC of the head and neck after failure of chemotherapy in patients treated with afatinib. Therefore, treatment of patients with these 2 conditions with afatinib is not experimental, and will follow conventional clinical management.

DETAILED DESCRIPTION:
Clinical objectives:

1. To determine the efficacy of afatinib in patients with germline MET-N375S polymorphism.
2. To determine the tolerability of afatinib in chemo-relapsed patients with germline MET-N375S polymorphism.

Research objectives:

1. To determine the prevalence of MET and TP53 mutations, as well as HER2 and MET amplification, in various cancers, particularly head and neck cancers and lung cancers.
2. To establish tumour cell lines, spheroids of xenografts for drug screening.

Endpoints of study:

1. To determine the response rate of SCC HN/lung with Met-N375S to afatinib.
2. The secondary endpoints include progression-free survival and toxicity.
3. Frequency of MET mutations and TP53 mutations in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be included in the study only if they meet all of the following criteria:

  1. Age 18 years or older
  2. Histologic or cytologic confirmation of metastatic squamous cell carcinoma of the lung or head and neck region, and has failed standard treatment.
  3. No other active malignancy within the past 24 months
  4. All subjects must have at least one tumour lesion (primary or metastatic) that is suitable for free-hand or image-guided biopsy at baseline.
  5. Clinical study will enroll patients genotyped positive for MET-N375S polymorphism.
  6. Eastern Cooperative Oncology Group (ECOG) performance status < 2
  7. Adequate organ function as defined by:

     a. Bone marrow function i. Haemoglobin ≥ 9g/dl ii. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L iii. Platelet count ≥ 75 x 109/L. b. Liver function i. Bilirubin < 2.5x upper limit of normal (ULN) ii. Alanine transaminase (ALT) and aspartate transaminase (AST) < 2.5x ULN or < 5x ULN if liver metastases are present iii. Prothrombin time (PT) within the normal range for the institution. c. Renal function i. Plasma creatinine <1.5x institutional ULN
  8. Capable of swallowing tablets
  9. Recovery from any previous drug- or procedure-related toxicity to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 Grade 0 or 1 (except alopecia), or to baseline preceding the prior treatment.
  10. Signed informed consent obtained before any study specific procedure. Subjects must be able to understand and be willing to sign the written informed consent.

Exclusion Criteria:

* 1. Chemotherapy, radiotherapy, surgery, immunotherapy or other therapy within 3 weeks of starting investigational medicinal product (IMP).

  2. Pregnancy or breastfeeding. 3. Women of childbearing potential not employing adequate contraception. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of study medication, and a negative result must be documented before start of study medication. Women of childbearing potential and men, must agree to use adequate contraception (barrier method of birth control) upon signing the informed consent form until at least 3 months after the last study drug administration 4. Known or suspected allergy to the investigational agent or any agent given in association with this study.

  5. Concurrent cancer which is distinct in primary site or histology from the cancer being evaluated in this study 6. Patients with CTCAE Grade 2 or higher peripheral neuropathy. 7. History of significant cardiac disease: congestive cardiac failure > NYHA class II, ongoing unstable angina, new-onset angina or myocardial infarction within the past 3 months

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
p-HER2 and p-MET status | 3 years
  using immunohistochemistry.
MET-N375S mRNA copy number | 3 years
  using RNAscope staining.
Identification of MET and TP53 mutations using droplet digital PCR (ddPCR) and Sanger sequencing. | 3 years
  DNA from the tumour specimens will be harvested for sequencing to identify cases with somatic mutations of TP53 gene. Changes in codon sequences will be reported.
  Germline DNA from the patients will be harvested from whole blood, and the polymorphic MET variant will be determined using ddPCR. Customised probes detecting wildtype MET allele or MET-N375S allele are designed to for genotyping (homozygous/heterozygous).
Presence of MET and HER2 amplification using fluorescence in situ hybridization (FISH) | 3 years
  FFPE samples retrieved from patients genotyped with MET-N375S polymorphism will be subjected to MET and HER2 testing Abbott PathVysion DNA test kits. Data will be analysed with fluorescence microscopy. HER2 amplification will be defined as gene copies versus chromosome 17 polysomy. MET amplification will be defined as gene copies per nucleus.
Interaction of cMet and HER2 receptor tyrosine kinases using proximity ligation assay (PLA) | 3 years
  PLA will be performed using DUOLINK in situ hybridization. Validation MET and HER2 antibodies will be used for the assay, and signal will be detected with fluorescence microscopy. Detection and quantification of positive signals will determine the presence of MET-HER2 interaction in clinical specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cancer Genome Atlas Research Network. Comprehensive genomic characterization of squamous cell lung cancers. Nature. 2012 Sep 27;489(7417):519-25. doi: 10.1038/nature11404. Epub 2012 Sep 9. PMID 22960745
- [Result] Liu Y, Zhang Q, Ren C, Ding Y, Jin G, Hu Z, Xu Y, Shen H. A germline variant N375S in MET and gastric cancer susceptibility in a Chinese population. J Biomed Res. 2012 Sep;26(5):315-8. doi: 10.7555/JBR.26.20110087. Epub 2012 Mar 29. PMID 23554766